CLINICAL TRIAL: NCT05909696
Title: Median Effective Dose of Rocuronium for the Prevention of Myofibrillation Caused by the Injection of Succinylcholine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20230610
Record Dates: First submitted 2023-06-10; First posted 2023-06-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Succinylcholine; Myofibrillation
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age range of 18 to 44 years olds (Experimental): Age range of 18 to 44 years olds The initial dose of rocuronium for pre-injection was set at 0.04mg/kg according to previous literature and preliminary test results. The dose of rocuronium was according to the patients' myofibrillation level. If there is no myofibrillation (negative reaction), the dose of rocuronium in the next patient will be reduced until the patient has myofibrillation. If there is myofibrillation (positive reaction), the dose of rocuronium will be increased in the next patient until the patient is no fibrillation.
  Interventions: Drug: rocuronium
- Age range of 45 to 59 years olds (Experimental): Age range of 18 to 44 years olds The initial dose of rocuronium for pre-injection was set at 0.04mg/kg according to previous literature and preliminary test results. The dose of rocuronium was according to the patients' myofibrillation level. If there is no myofibrillation (negative reaction), the dose of rocuronium in the next patient will be reduced until the patient has myofibrillation. If there is myofibrillation (positive reaction), the dose of rocuronium will be increased in the next patient until the patient is no fibrillation.
  Interventions: Drug: rocuronium
- Age range of 60 to 80 years olds (Experimental): Age range of 18 to 44 years olds The initial dose of rocuronium for pre-injection was set at 0.04mg/kg according to previous literature and preliminary test results. The dose of rocuronium was according to the patients' myofibrillation level. If there is no myofibrillation (negative reaction), the dose of rocuronium in the next patient will be reduced until the patient has myofibrillation. If there is myofibrillation (positive reaction), the dose of rocuronium will be increased in the next patient until the patient is no fibrillation.
  Interventions: Drug: rocuronium

INTERVENTIONS:
Drug: rocuronium — Advanced intravenous injection of rocuronium before the succinylcholine injection

SUMMARY:
Succinylcholine is an important component of rapid sequential induction of general anesthesia because of its rapid onset and short duration of action. However, myofibrillation is a common complication after succinylcholine injection and may lead to persistent postoperative myalgia, increased intraocular, intragastric and intracranial pressure in patients. Increased risk of peri-induction and postoperative patient discomfort. The effectiveness of rocuronium bromide pretreatment in reducing succinylcholine-induced myalgias has been demonstrated in several recent studies. However, the half effective amount of rocuronium pretreatment for small doses is not well known. Therefore, this study applied the Dixon sequential method to investigate the ED50 of preemptive intravenous rocuronium bromide for the prevention of succinylcholine-induced myofibrillation and to investigate the effect of age factor on the ED50 of rocuronium bromide for the prevention of succinylcholine-induced myofibrillation to provide a reference for the rational clinical selection of rocuronium bromide dose.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ranged from 18 to 80.
2. ASA grade I-II

Exclusion Criteria:

1. Possible airway difficulties,
2. allergies or contraindications to rocuronium and succincholine ，
3. cardiac insufficiency,
4. hepatic or renal dysfunction,
5. neuromuscular disease,
6. surgery lasting more than 2 hours,
7. taking any known drug that has interaction with neuromuscular blockers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The appearance of myofibrillation | Average 45 seconds
  Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tian S, Chen C, Wang S, Feng S, Wang M, Liu X, Bao T, Zhang Z. Median effective dose of rocuronium for the prevention of succinylcholine-induced fasciculation: an age-stratified study. BMC Anesthesiol. 2025 Dec 10;26(1):35. doi: 10.1186/s12871-025-03546-5. PMID 41366298